CLINICAL TRIAL: NCT00002995
Title: Actinomycin D and Vincristine With or Without Radiation Therapy, for Newly Diagnosed Patients With Low-Risk Rhabdomyosarcoma or Undifferentiated Sarcoma: IRS-V Protocol
Brief Title: Combination Chemotherapy With or Without Radiation Therapy in Treating Patients With Newly Diagnosed Rhabdomyosarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: D9602; COG-D9602 (Other: Children's Oncology Group); CCG-D9602 (Other: Children's Cancer Group); POG-D9602 (Other: Pediatric Oncology Group); IRS-D9602 (Other: Intergroup Rhabdosarcoma); CDR0000065542 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Sarcoma
Keywords: embryonal childhood rhabdomyosarcoma; embryonal-botryoid childhood rhabdomyosarcoma; previously untreated childhood rhabdomyosarcoma; adult rhabdomyosarcoma; adult malignant mesenchymoma; childhood malignant mesenchymoma; nonmetastatic childhood soft tissue sarcoma; stage II adult soft tissue sarcoma; stage III adult soft tissue sarcoma; stage I adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Rhabdomyosarcoma; Malignant mesenchymal tumor | interventions — Dactinomycin; Filgrastim; sargramostim; Cyclophosphamide; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: dactinomycin
Biological: filgrastim
Biological: sargramostim
Drug: cyclophosphamide
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known whether chemotherapy is more effective with or without radiation therapy in treating patients who have rhabdomyosarcoma.

PURPOSE: Phase III trial to compare the effectiveness of chemotherapy with or without radiation therapy in treating patients who have newly-diagnosed rhabdomyosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the failure-free survival (FFS) rate in patients with newly diagnosed low-risk rhabdomyosarcoma of embryonal or botryoid subtype meeting criteria for group I after treatment with dactinomycin and vincristine with or without radiotherapy.
* Determine the FFS rate in these patients meeting criteria for group II after treatment with dactinomycin, vincristine, and cyclophosphamide with or without radiotherapy.
* Determine the FFS rate in patients with ectomesenchymomas containing rhabdomyosarcomatous elements (embryonal histiotype) who receive one of the above treatments.
* Determine new molecular markers specific to embryonal and botryoid tumor histologies which are of diagnostic and prognostic significance in patients treated with these regimens.

OUTLINE: Patients are assigned to 1 of 2 groups, depending on histology and site of disease.

* Group I (favorable tumor site, negative lymph nodes, stage 1, clinical group I, IIA, or III (orbit only), node negative [N0] OR unfavorable tumor site, negative or unknown lymph nodes, stage 2, clinical group I): Patients receive vincristine IV over 1 minute weekly for 8 weeks and dactinomycin IV over 1 minute once every 3 weeks for 4 doses. Treatment repeats every 12 weeks for 4 courses. Radiotherapy is administered to patients with clinical group II or III disease on weeks 3-8.
* Group II (favorable tumor site, positive lymph nodes, stage 1, clinical group III (orbit only), node positive [N1] OR favorable tumor site except orbit, any lymph nodes, stage 1, clinical group III OR unfavorable tumor site, stage 2, clinical group II OR unfavorable tumor site, stage 3, clinical group I or II): Patients receive vincristine and dactinomycin as in group I. Patients also receive cyclophosphamide IV over 30-60 minutes and filgrastim (G-CSF) or sargramostim (GM-CSF) subcutaneously once daily beginning 24 hours after completion of chemotherapy and continuing for 10 days or until blood counts recover. Radiotherapy is administered on weeks 3-8, 12-17, or 28-33, if clinically indicated as in group I.

Patients are followed every 3-4 months for 3 years (4 years after diagnosis), every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 254 patients for group I will be accrued for this study within 6 years. Approximately 12 patients per year will be accrued for group II.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed embryonal (EMB) rhabdomyosarcoma (RMS) or botryoid or spindle cell variants of EMB RMS or embryonal ectomesenchymoma meeting 1 of the following criteria:

  * Stage 1, no clinical group IV: Tumor in favorable site (orbit, head and neck [excluding parameningeal], genitourinary [not bladder/prostate], or biliary tract) and no metastatic disease
  * Stage 2 or 3, clinical group I or II: Tumor in unfavorable site (bladder/prostate, extremity, cranial parameningeal, trunk, retroperitoneum, pelvis, perineal/perianal, intrathoracic, gastrointestinal, or liver), no gross residual disease after initial surgery, and no metastatic disease
* Must have ipsilateral lymph node dissection if age 10 or over with primary paratesticular cancer OR under age 10 with clinically positive regional lymph nodes
* Low risk of recurrence
* Previously untreated disease
* No alveolar RMS or undifferentiated sarcoma
* No intermediate-risk disease
* No metastatic disease at diagnosis

PATIENT CHARACTERISTICS:

Age:

* Under 50

Performance status:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin elevation secondary to biliary or hepatic primaries allowed

Renal:

* Creatinine elevation secondary to tumor obstruction allowed

Other:

* No uncontrolled infection
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Max Age: 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 483 (Actual)
Dates: Start 1997-08; Primary Completion 2006-09 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Failure-free survival

CONTACTS AND LOCATIONS:
Overall Officials: R. Beverly Raney, MD, Study Chair — M.D. Anderson Cancer Center
Locations (233):
- United States (205):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - University of South Alabama Cancer Research Institute, Mobile, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center/Kaiser Foundation Hospital - San Diego, San Diego, California
  - Children's Hospital and Health Center, San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Children's Hospital of Denver, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - University of Connecticut Comprehensive Cancer Center at University of Connecticut Health Center, Farmington, Connecticut
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Shands Cancer Center at the University of Florida Health Science Center, Gainesville, Florida
  - Joe DiMaggio Children's Hospital at Memorial, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Nemours Children's Clinic-Orlando, Orlando, Florida
  - Sacred Heart Children's Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Children's Hospital, Tampa, Florida
  - St. Mary's Hospital, West Palm Beach, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Scottish Rite Campus, Atlanta, Georgia
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Mountain States Tumor Institute - Boise, Boise, Idaho
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois Medical Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Children Cancer Center at Riley Hospital for Children, Indianapolis, Indiana
  - St. Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Wesley Medical Center, Wichita, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Baystate Regional Cancer Program at Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health and DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - William Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Children's Hospitals and Clinics - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Hospitals and Clinics - Minnesota, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Omaha, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey at Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Valerie Fund Children's Center at Atlantic Health, Summit, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - Comprehensive Cancer Center at Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - University Hospital at State University of New York - Upstate Medical University, Syracuse, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospitals, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Leo W. Jenkins Cancer Center of University Health Systems of Eastern Carolina, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Dakota Cancer Institute at Innovis Health - Dakota Clinic, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Forum Health-Tod Childrens Hospital, Youngstown, Ohio
  - Children's Hospital at Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Doernbecher Children's Hospital at Oregon Health & Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sioux Valley Hospital at University of South Dakota Medical Center, Sioux Falls, South Dakota
  - East Tennessee State University Cancer Center at Johnson City Medical Center, Johnson City, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Children's Hospital of Austin, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MBCCOP - South Texas Pediatrics, San Antonio, Texas
  - Methodist Cancer Center at Methodist Specialty and Transplant Hospital, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Center for Cancer Prevention and Care at Scott and White Clinic, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Carilion Medical Center for Children, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Cabell Huntington Hospital, Huntington, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (6):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (15):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre de Recherche du Centre Hospitalier de l'Universite Laval, Sainte-Foy, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- Starship Children's Hospital, Auckland, New Zealand
- Puerto Rico (2):
  - Puerto Rico Cancer Center at University of Puerto Rico - Medical Sciences Campus, San Juan
  - San Jorge Childrens Hospital, Santurce
- Switzerland (3):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva
  - Swiss Pediatric Oncology Group Lausanne, Lausanne

REFERENCES:
- [Background] Malempati S, Rodeberg DA, Donaldson SS, Lyden ER, Anderson JR, Hawkins DS, Arndt CA. Rhabdomyosarcoma in infants younger than 1 year: a report from the Children's Oncology Group. Cancer. 2011 Aug 1;117(15):3493-501. doi: 10.1002/cncr.25887. Epub 2011 Jan 24. PMID 21264837
- [Background] Walterhouse DO, Meza JL, Breneman JC, Donaldson SS, Hayes-Jordan A, Pappo AS, Arndt C, Raney RB, Meyer WH, Hawkins DS. Local control and outcome in children with localized vaginal rhabdomyosarcoma: a report from the Soft Tissue Sarcoma committee of the Children's Oncology Group. Pediatr Blood Cancer. 2011 Jul 15;57(1):76-83. doi: 10.1002/pbc.22928. Epub 2011 Feb 4. PMID 21298768
- [Result] Breneman J, Meza J, Donaldson SS, Raney RB, Wolden S, Michalski J, Laurie F, Rodeberg DA, Meyer W, Walterhouse D, Hawkins DS. Local control with reduced-dose radiotherapy for low-risk rhabdomyosarcoma: a report from the Children's Oncology Group D9602 study. Int J Radiat Oncol Biol Phys. 2012 Jun 1;83(2):720-6. doi: 10.1016/j.ijrobp.2011.06.2011. Epub 2011 Nov 19. PMID 22104356
- [Result] Raney RB, Walterhouse DO, Meza JL, Andrassy RJ, Breneman JC, Crist WM, Maurer HM, Meyer WH, Parham DM, Anderson JR. Results of the Intergroup Rhabdomyosarcoma Study Group D9602 protocol, using vincristine and dactinomycin with or without cyclophosphamide and radiation therapy, for newly diagnosed patients with low-risk embryonal rhabdomyosarcoma: a report from the Soft Tissue Sarcoma Committee of the Children's Oncology Group. J Clin Oncol. 2011 Apr 1;29(10):1312-8. doi: 10.1200/JCO.2010.30.4469. Epub 2011 Feb 28. PMID 21357783